CLINICAL TRIAL: NCT06143215
Title: Clinical Efficacy of Different Revision Times in the Reulceration Rate in Persons with Diabetes and Remission: a Three Arm Double Blind Randomized Clinical Trial
Brief Title: Clinical Efficacy of Different Revision Times in the Reulceration Rate in Persons with Diabetes and Remission
Acronym: Diatime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Mateo López-Moral, DPM, PhD, Prof. Dr, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Diatime_061123
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot; Reulceration; Prevention
MeSH Terms: conditions — Diabetic Foot | interventions — Second-Look Surgery

STUDY DESIGN:
Intervention Model Description: Three arms parallel randomized clinical trial
Masking Description: No masking is possible to be performed in the planned RCT due to the nature of the intervention (time dependent).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fourweeks revision group (Experimental): Patients will be clinically revised in a 4-weeks basis
  Interventions: Behavioral: 4 weeks revision
- Eightweeks revision group (Active Comparator): Patients will be clinically revised in a 8-weeks basis
  Interventions: Behavioral: 4 weeks revision
- Twelveweeks revision group (Experimental): Patients will be clinically revised in a 12-weeks basis
  Interventions: Behavioral: 4 weeks revision

INTERVENTIONS:
Behavioral: 4 weeks revision — In the literature is described to clinically revise patients in a 4-6 weeks basis, despite this expert recommendation, no previous research has clinically evaluated if 4-8-12 weeks revision times could change diabetic foot reulceration rate.

SUMMARY:
The goal of this three arms randomized clinical trial is to compare different revision times in persons with diabetes at high risk of suffering a diabetic foot reulceration (patients in remission). The literature suggests to clinically check the patients in a 4-12 weeks basis, despite this, this recommendation is based in expert opinions.

The main question it aims to answer is:

- Does different revision times could affect the reulceration rate in persons with diabetes in remission. Different revision time will be 2 weeks, 4 weeks and 6 weeks.

DETAILED DESCRIPTION:
The planned RCT try to elucidate if there exist any difference in ulcer recurrence between different revisions times in persons with a previous healed diabetic foot ulcer and currently under remission.

There will exist three different groups for analyses after randomization:

* Group 1: patients revised every fourweeks.
* Group 2: patients revised every eightweeks.
* Group 3: patients revised every twelveweeks.

Main outcome measure will include:

- Recurrence: the outcome measure was based on recurrent events in the foot in a binary basis (patient with a recurrent event or patient without a recurrent event), as defined according to the IWGDF guidelines. Recurrent events were considered as breaks in the foot skin at the epidermis and part of the dermis level.

Secondary outcome measure will include:

* Minor lesions: defined as non ulcerative lesions of the skin on the plantar aspect of the foot and included abundant callus, hemorrhage, or a blister.
* Minor amputations: evaluated in a monthly basis during the 1-year prospective period

Follow-up period: all the sample will be followed-up depending on the randomization group up to a 1-year prospective period. In every visit de principal investigator will perform debridement of high-risk points, such as minor lesions or calluses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Type 1 or type 2 diabetes.
* Presence of diabetic polyneuropathy (diagnosed as an inability to sense the pressure of a 10-g Semmes-Weinstein monofilament at three plantar foot sites and/or a vibration perception threshold >25 V, as assessed using a bio-tensiometer.
* Patients classified as high-risk patients (risk 3 patients according to the IWGDF guidance). Previous healed diabetic foot ulcer.

Exclusion Criteria:

* Active diabetic foot ulcers during inclusion.
* Active Charcot foot process.
* Conditions other than diabetes also associated with foot ulcers were excluded from the study as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | From randomization to first documented diabetic foot ulcer appearance, assessed up to 48 weeks.
  Defined as as break in the foot skin at the epidermis and part of the dermis level.

SECONDARY OUTCOMES:
Minor lesion rate | From randomization to first documented diabetic foot ulcer appearance, assessed up to 48 weeks.
  Defined as non ulcerative lesions of the skin on the plantar aspect of the foot and included abundant callus, hemorrhage, or a blister.
Minor amputation rate | From randomization to first documented diabetic foot ulcer appearance, assessed up to 48 weeks.
  Need for minor amputation secondary to ulcer recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria de Podología de la Universidad Complutense de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Moral M, Garcia-Madrid M, Garcia-Morales E, Garcia-Alvarez Y, Alvaro-Afonso FJ, Lazaro-Martinez JL. Comparison of 4, 8, and 12 week screening and foot care frequencies in persons in remission: The DIATIME comparative efficacy study - A randomized clinical trial. Diabetes Res Clin Pract. 2025 Dec;230:112962. doi: 10.1016/j.diabres.2025.112962. Epub 2025 Oct 24. PMID 41139025